CLINICAL TRIAL: NCT06887829
Title: The Randomized Clinical Trial of Low-Dose Radiotherapy for Knee Osteoarthritis
Brief Title: Radio- KO Radiotherapy for Knee Osteoarthritis Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Stephen P. Merry, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 24-006759
Record Dates: First submitted 2025-03-07; First posted 2025-03-20 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Low dose radiotherapy (Active Comparator): Low dose radiation therapy for knee osteoarthritis
  Interventions: Radiation: Low dose radiotherapy
- Placebo (Sham Comparator): No radiation therapy
  Interventions: Other: Sham comparator

INTERVENTIONS:
Radiation: Low dose radiotherapy — Participants will receive low dose radiotherapy (0.5 Gy) 3 times per week, for two weeks delivered via the X-Strahl Orthovoltage device.
  Arms: Low dose radiotherapy
Other: Sham comparator — Participants will receive identical treatment 3 times per week, for two weeks delivered via the X-Strahl Orthovoltage device, without radiation.
  Arms: Placebo

SUMMARY:
The primary aim of this study is to investigate whether low-dose radiotherapy is an effective treatment to reduce the pain of knee osteoarthritis. A secondary aim is to determine whether patients experience any more measurable side effects than those receiving sham treatments.

DETAILED DESCRIPTION:
This single center, single-blinded, sham-controlled randomized controlled trial will compare low dose radiation therapy and sham radiation therapy for knee osteoarthritis. Participants with symptomatic knee OA based on clinical and radiographic criteria will be randomized 1:1 to receive 0.5 Gy LDRT over 2 weeks ideally on a Monday-Wednesday-Friday three times each week for two weeks treatment course for a total of 3 Gray or identical sham treatment (an identical procedure without the radiation). Non-responders to the initial Low-Dose Radiotherapy (LDRT)/sham treatment will receive a second treatment course of 0.5 Gy Low-Dose Radiotherapy (LDRT) or sham repeat treatment course over 2 weeks x 6 depending on their randomization (treatment arm participants receiving a second treatment course and sham arm participants receiving a second course of identical sham treatments without radiation). Intermittent and Constant Osteoarthritis Pain (ICOAP) outcome scales will be emailed to all participants for completion at baseline and weekly for six months. The study will thus terminate after all participants have completed 6 months of time in the study.

ELIGIBILITY:
Inclusion Criteria:

* age 50-85 years

  * ICOAP pain scale A1 at least moderate intensity or B6 at least moderate intensity
  * diagnosed with primary knee OA ICD-10 codes M17.x
  * history of morning stiffness in knees that lasts less than 30 minutes
  * history of crepitus without a history of warmth, redness or sudden onset of swelling
  * physical exam findings of medial or lateral joint line tenderness on palpation that is in the same location as the knee pain for which their primary care provider has ordered an intraarticular steroid injection into the same knee.
  * absence of primary knee pain in the pes anserine or hamstring or gastrocnemius tendons
  * radiographic Kellgren-Lawrence grade 2-3 on 4-view knee x-rays taken within the last year
  * ability to complete surveys in English

Exclusion Criteria:

* Kellgren-Lawrence grade 1 or 4

  * pregnancy or women 54 years and younger with potential for pregnancy (if they or their partner have not had tubal ligation, hysterectomy, or vasectomy)
  * history of ipsilateral intraarticular knee surgery
  * use of injected corticosteroids within 3 months or hyaluronans within 6 months or within 1 month if there was no sustained improvement post-injection of either corticosteroid or hyaluronan.
  * history of trauma to this knee in the last year that clearly caused the pain now present
  * history of RA, gout, pseudogout, hemarthroses (eg, hemophilic arthropathy) or other inflammatory arthritis involving this knee
  * history of symptomatic hip OA
  * history of psychosis, personality disorder, uncontrolled affective disorder
  * history of fibromyalgia
  * malignancy requiring active treatment
  * current regular use of opiate analgesics, PRP, or acupuncture for the knees

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-06-04 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Change in Area Under the Curve (AUC) of ICOAP Scores | Baseline, 6 months
  Change in the Intermittent and Constant Osteoarthritis Pain (ICOAP) outcome scale weekly for six months after intervention analyzed as area under the curve of patients with Kellgren-Lawrence grade 2-3 knee OA.
Analgesic use frequency in treatment vs. sham participants | 6 months
  Differences in the rate of improvement between the 2 groups with analysis to include time points of 2 months and 4 months after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P. Merry, M.D., Principal Investigator — Mayo Clinic; Paul D. Brown, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No